CLINICAL TRIAL: NCT04695756
Title: Impact of Coronavirus Disease 2019 (COVID-19) Epidemic in Patients Requiring Liver Transplantation
Brief Title: Liver Transplantation and Coronavirus Disease 2019 (COVID-19)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: National Agency for Scientific and Technological Promotion, Argentina (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, PhD, MPH, MD, Coordinator of the non-sponsored area of the departemt of Research, Hospital Italiano de Buenos Aires
Other Study IDs: 1405
Record Dates: First submitted 2021-01-04; First posted 2021-01-05 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Liver Transplant
MeSH Terms: conditions — COVID-19 | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People who require liver transplant: We will compare the year before the beginning of the COVID-19 Pandemia with the period during the COVID-19 Pandemia.
  Interventions: Other: COVID-19 pandemic

INTERVENTIONS:
Other: COVID-19 pandemic — The exposure of this observational study is the COVID-19 pandemic

SUMMARY:
The COVID-19 pandemic together with the strategies that are applied to control it are generating high morbidity and mortality worldwide. Its impact on health systems is worrisome, affecting all the population, even those who are not infected or at risk.

The indirect impact of the COVID-19 pandemic on the access to the medical care of patients on the waiting list for organ transplantation might be multifactorial, including the need to relocate health-related resources (medical personnel, supplies, critical care unit beds, etc), the risk of COVID-19 transmission among donors or patients on the waiting list, and also after transplantation. Additionally, the pandemic reduces significantly the donor pool.

We consider that it is important to assess the impact that the pandemic has in particular individual populations, such as in patients requiring a liver transplant. Along with the lockdown, the rate of organ donation has dropped, and liver transplant programs across the world have reduced or suspended their activity. Unfortunately, this is invariably associated with an increase in mortality on the waiting list.

Knowing the impact of the pandemic on patients who require a liver transplant will provide tools to understand and plan the health resources related to the care of these patients, not only at present but also in the following years.

DETAILED DESCRIPTION:
The COVID-19 pandemic together with the strategies that are applied to control it is generating high morbidity and mortality worldwide. Its impact on health systems is worrisome, affecting all the population, even those who are not infected or at risk.

The indirect impact of the COVID-19 pandemic on the access to the medical care of patients on the waiting list for organ transplantation might be multifactorial, including the need to relocate health-related resources (medical personnel, supplies, critical care unit beds, etc), the risk of COVID-19 transmission among donors or patients on the waiting list, and also after transplantation. Additionally, the pandemic reduces significantly the donor pool.

We consider that it is important to assess the impact that the pandemic has in particular individual populations, such as in patients requiring a liver transplant. Along with the lockdown, the rate of organ donation has dropped, and liver transplant programs across the world have reduced or suspended their activity. Unfortunately, this is invariably associated with an increase in mortality on the waiting list.

Knowing the impact of the pandemic on patients who require a liver transplant will provide tools to understand and plan the health resources related to the care of these patients, not only at present but also in the following years.

The primary objectives of the study will be

To Compare the following outcomes in patients requiring liver transplantation during the epidemiological weeks of COVID-19 pandemic in Argentina and the same weeks of 2019 according to national data registry of procurement and transplantation:

1. Number of patients registered on the liver transplant waiting list
2. Number of deaths on the liver transplant waiting list
3. Number of liver transplants

For this purpose, we will carry out a time series analyses using the national data registry of procurement and transplantation database. The effect of both periods will be analysed as time interrupted series, which is a quasi-experimental design. The following two periods will be compared as segments of the interrupted time series:

* Baseline period (Period not exposed to the pandemic represented by the same epidemiological weeks of 2019 )
* Pandemic period COVID-19. (Period between the epidemiological weeks of 2020 affected by the pandemic declared by the WHO from 11/March/2020)

The unit of analysis will be the epidemiological weeks, and the study population will be all Argentinian over 17 years of age. Regarding patients who require liver transplantation, those who registered for isolated liver transplantation in the National Procurement and Transplant Institute will be included.

A Poisson regression model will be used to assess the association between the period and the incidence of the events of interest. ARIMA models will be used following the 4 steps proposed by Box and Jenkings

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years-old
* Argentinean

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a population-based study. The study population is the Argentine population.
  Regarding the patients, those who are registered on the national waiting list for isolated liver transplantation will be included.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
To compare the number of patients registered on the liver transplant waiting list during the epidemiological weeks of COVID-19 pandemic in Argentina and the same weeks of 2019 according to national data registry of procurement and transplantation | 1 year
  During the study period, patients who are registered on the transplant waiting list will be included. The data source will be the national transplant database.

SECONDARY OUTCOMES:
To compare the number of deaths on the liver transplant waiting list during the epidemiological weeks of COVID-19 pandemic in Argentina and the same weeks of 2019 according to national data registry of procurement and transplantation | 1 year
  During the study period, patients who die on the transplant waiting list will be registered. The data source will be the national transplant database.
To compare the number of liver transplants during the epidemiological weeks of COVID-19 pandemic in Argentina and the same weeks of 2019 according to national data registry of procurement and transplantation | 1 year
  During the study period, the number of liver transplants who are performed will be registered. The data source will be the national transplant database.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastián Marciano, MS, Msc, Study Chair — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No